CLINICAL TRIAL: NCT07246148
Title: A Randomized Controlled Trial on Non-Invasive Continuous Blood Pressure Monitoring as an Alternative to Radial Arterial Catheterization in Patients Undergoing Coil Embolization for Intracranial Aneurysms
Brief Title: NOn-inVAsive Blood Pressure Monitoring in Intracranial Aneurysm Embolization
Acronym: NOVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, JangHun Kim, Principal Investigator, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: K2025-2494-001
Record Dates: First submitted 2025-10-01; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Aneurysms; Intracranial Aneurysms; Coil Embolization; Hemodynamic Instability; Noninvasive Cardiac Monitoring
Keywords: non-invasive blood pressure monitoring; continuous arterial blood pressure monitoring; coil embolization; neuroanesthesia; cerebral oximetry; radial arterial catheterization
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio into two parallel groups: the experimental arm (non-invasive blood pressure monitoring using ClearSight system) and the control arm (invasive radial arterial catheter monitoring).
Who Masked: Outcomes Assessor
Masking Description: This study is conducted as a partial double-blind trial. Patients cannot be blinded to the presence or absence of a radial arterial catheter after the procedure. The anesthesiologist managing hemodynamics is also not blinded due to the differences in monitoring displays. However, the neurosurgeon performing the coil embolization, who does not have access to hemodynamic monitoring screens, remains blinded to group allocation. Outcome assessors and statisticians are fully blinded, and all event adjudications will be conducted using predefined criteria and de-identified datasets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NVBP group (Experimental): Participants undergo continuous non-invasive blood pressure (NVBP) monitoring using the ClearSight system (Edwards Lifesciences, Irvine, CA, USA) during coil embolization for intracranial aneurysm. Cerebral oxygen saturation is simultaneously monitored with O₃® Regional Oximetry (Masimo, CA, USA). A femoral arterial catheter placed for endovascular access may serve as a backup for safety, but invasive radial arterial catheterization is not performed.
  Interventions: Device: Non-invasive continuous blood pressure monitoring
- IABP group (Active Comparator): Participants undergo standard invasive arterial blood pressure (IABP) monitoring via radial arterial catheterization during coil embolization. Cerebral oxygen saturation is also monitored with O₃® Regional Oximetry (Masimo, CA, USA), identical to the NVBP group.
  Interventions: Device: Invasive arterial blood pressure monitoring

INTERVENTIONS:
Device: Non-invasive continuous blood pressure monitoring — Continuous arterial blood pressure monitoring using a finger-cuff technology (e.g., ClearSight system). Applied in the experimental NVBP group.
  Arms: NVBP group
Device: Invasive arterial blood pressure monitoring — Standard radial arterial catheterization for continuous invasive blood pressure monitoring. Applied in the IABP control group.
  Arms: IABP group

SUMMARY:
The goal of this clinical trial is to evaluate whether non-invasive continuous blood pressure monitoring (NVBP) using the ClearSight system can safely serve as an alternative to radial arterial catheterization for invasive arterial blood pressure monitoring (IABP) in patients undergoing coil embolization for unruptured intracranial aneurysms.

The main questions it aims to answer are:

* Does NVBP monitoring detect intraoperative hypotension and hypertension events with similar reliability compared to IABP?
* Does NVBP monitoring reduce the need for invasive arterial catheterization without compromising patient safety or clinical outcomes?

Researchers will compare patients assigned to NVBP monitoring with those receiving conventional IABP monitoring.

Participants will:

* Be randomly assigned to NVBP monitoring or standard IABP monitoring during coil embolization.
* Receive continuous monitoring of cerebral oxygenation with near-infrared spectroscopy (rSO₂).
* Undergo standard anesthesia induction, maintenance, and postoperative intensive care protocols.
* Have their intraoperative hemodynamic events, vasopressor use, and postoperative outcomes recorded up to 30 days after the procedure.

DETAILED DESCRIPTION:
Intracranial aneurysm coil embolization is a widely accepted treatment for unruptured aneurysms, but the procedure is frequently accompanied by hemodynamic instability, particularly episodes of hypotension and hypertension, which may increase the risk of neurological or cardiovascular complications. Continuous and reliable arterial blood pressure monitoring is therefore critical during the periprocedural period.

The conventional standard of care has been invasive arterial blood pressure (IABP) monitoring using a radial arterial catheter. Although IABP provides accurate real-time hemodynamic data, it is associated with procedural risks such as bleeding, hematoma, arterial occlusion, distal ischemia, infection, and patient discomfort. These risks are particularly relevant in patients undergoing neuroendovascular procedures where vascular access and anticoagulation may already increase complication risk.

The ClearSight™ system (Edwards Lifesciences, Irvine, CA, USA) is a non-invasive continuous blood pressure monitoring device that uses a finger cuff based on the volume clamp method and pulse contour analysis. Previous studies have validated its use in a variety of surgical and perioperative settings, including obese patients, vascular surgery, and cardiac surgery [Kim et al., 2014; Maheshwari et al., 2018; Bugarini et al., 2021; Chapalain et al., 2024]. However, its role as a primary monitoring modality during neuroendovascular procedures has not been fully established.

This randomized controlled trial (NOVA study) is designed to determine whether non-invasive continuous blood pressure monitoring (NVBP) can serve as a safe and effective alternative to radial IABP in patients undergoing coil embolization for unruptured intracranial aneurysms. Patients will be randomized in a 1:1 ratio to receive either NVBP monitoring (experimental arm) or standard IABP monitoring (control arm). All participants will also undergo cerebral oxygenation monitoring with O₃® Regional Oximetry (Masimo, CA, USA) to detect potential cerebral desaturation events.

In the NVBP group, invasive arterial pressure will not be obtained from a radial catheter but may be secondarily recorded from a femoral arterial catheter used for the endovascular procedure itself. Importantly, the femoral arterial waveform will not be displayed to the anesthesiologist but will be recorded by nursing staff to ensure patient safety and allow for event adjudication if NVBP and IABP values diverge significantly.

The primary endpoint of this study is the intraoperative incidence of hemodynamic events, defined as episodes of hypotension (mean arterial pressure <65 mmHg sustained for ≥1 minute) or hypertension (systolic blood pressure >120 mmHg sustained for ≥1 minute). Secondary endpoints include vasopressor and antihypertensive drug use (type, dose, frequency), incidence of cerebral desaturation events (≥20% reduction from baseline or absolute rSO₂ <50), ICU admission and length of stay, overall hospital length of stay, 30-day mortality, reoperation rate, and incidence of major postoperative complications (neurologic, cardiovascular, or acute kidney injury).

To minimize performance bias, intraoperative management will follow a standardized anesthetic protocol including induction with propofol, rocuronium, and remifentanil; maintenance with sevoflurane (1 MAC); ventilation targeting normocapnia; and postoperative reversal and extubation criteria. Clinical decision-making for vasoactive drug administration will follow predefined thresholds based on both blood pressure and rSO₂ monitoring criteria.

This study aims to provide pilot-level evidence on whether NVBP can reduce the need for radial arterial catheterization without compromising intraoperative safety or postoperative outcomes. If successful, NVBP may represent a less invasive, safer, and patient-friendly monitoring option for neurointerventional procedures, with broader implications for perioperative practice in patients where invasive arterial access is either undesirable or technically challenging.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥19 and ≤80 years old) scheduled for elective coil embolization of unruptured intracranial aneurysms under general anesthesia.
* American Society of Anesthesiologists (ASA) physical status classification I-III.

Exclusion Criteria:

* Patients who do not provide informed consent.
* Patients unable to understand or follow study instructions due to physical or mental limitations.
* Patients in whom radial arterial catheterization is not feasible (e.g., peripheral vascular disease, skin disorders at the insertion site, absence of radial/ulnar artery, or orthopedic conditions of the upper extremity).
* Patients with peripheral vascular circulatory disorders.
* Patients with morbid obesity (BMI ≥ 40 kg/m²) [Eley et al., 2021].
* Patients who are hemodynamically unstable preoperatively or expected to be unstable during the perioperative period.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Intra-procedural hemodynamic instability events (hypotension or hypertension events) | During the procedure (Day 0)
  Incidence of hemodynamic instability during coil embolization. Hypotension is defined as mean arterial pressure (MAP) < 65 mmHg sustained for ≥ 1 minute. Hypertension is defined as systolic arterial pressure > 120 mmHg sustained for ≥ 1 minute.

SECONDARY OUTCOMES:
Use of vasoactive medications | During the procedure (Day 0)
  Name of vasoactive medications (vasopressors or antihypertensives) administered during the procedure
Dose of vasoactive medications (vasopressors or antihypertensives) | During the procedure (Day 0)
  cumulative dose of vasoactive medications administered during the procedure.
Cerebral oxygen desaturation events | During the procedure (Day 0)
  Incidence of cerebral oxygen desaturation, defined as ≥20% decrease from baseline or an absolute value <50 for ≥1 minute, measured by near-infrared spectroscopy (NIRS).
Length of hospital stay | Discharge day (typically postoperative 2 - 14 days)
  Duration (day) of hospitalization after coil embolization until discharge.
Incidence of ICU admission | Discharge day (typically postoperative 2 - 7 days)
  Incidence of ICU admission after embolization between two groups
length of stay in ICU | Discharge day (typically postoperative 2 - 7 days)
  duration of ICU stay (day)
30-day mortality | Postoperative Day 30
  All-cause mortality within 30 days after the procedure.
Major complications within 30 days | Postoperative Day 30
  Incidence of neurological complications, cardiovascular complications, and acute kidney injury (KDIGO criteria).
Event detection rate of NVBP vs IABP | Postoperative Day 30
  Comparison of the ability of non-invasive blood pressure monitoring vs invasive arterial blood pressure monitoring to detect hypotension, hypertension, or cerebral desaturation events.

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hoon Kim, M.D., Ph.D., Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
The plan for IPD sharing has not been finalized. Although de-identified data may be valuable for future research, the study is investigator-initiated at a single center and does not currently have a secure platform for external data sharing. Data sharing may be reconsidered in the future after publication, depending on institutional policies and available resources.